CLINICAL TRIAL: NCT00128830
Title: An Open-Label Trial With TMC125 in HIV-1 Infected Subjects, Who Were Randomized to a TMC125 Treatment Arm in a Sponsor-Selected TMC125 Trial and Were Treated for at Least 48 Weeks
Brief Title: A Study With TMC125 in Human Immunodeficiency Virus (HIV) Type 1 Infected Patients, Who Were Treated With TMC125 Arm in a Sponsor-Selected TMC125 Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR002731; TMC125-C229 (Other: Tibotec Pharmaceuticals, Ireland); NCT00980772 (obsolete NCT alias)
Record Dates: First submitted 2005-08-08; First posted 2005-08-10 (Estimated); Results first posted 2013-04-09 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Human Immunodeficiency Virus Type 1
Keywords: Human Immunodeficiency Virus Type 1; HIV-1 infection; TMC125; Etravirine; Enfuvirtide; Antiretroviral therapy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — etravirine; Protease Inhibitors; Enfuvirtide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Etravirine + 2 antiretrovirals (Experimental)
  Interventions: Drug: Etravirine (ETR); Drug: Nucleotide reverse transcriptase inhibitors (NRTIs); Drug: Protease inhibitors (PIs); Drug: Enfuvirtide (ENF)

INTERVENTIONS:
Drug: Etravirine (ETR) — Participants will receive 800 mg of ETR (2 x 4 tablets of formulation TF035) twice daily and after the formulation switch they will receive 200 mg of ETR (2 x 2 tablets of formulation F060) twice daily until the participants benefitted from etravirine or it became comercially available.
  Other Names: TMC125
Drug: Nucleotide reverse transcriptase inhibitors (NRTIs) — Participants will receive 2 additonal approved antiretrovirals (ARVs) along with ETR. ARVs may be NRTIs and/or allowed protease inhibitors (PIs) and/or enfuvirtide (ENF).
Drug: Protease inhibitors (PIs) — Participants will receive 2 additonal approved antiretrovirals (ARVs) along with ETR. ARVs may be NRTIs and/or allowed protease inhibitors (PIs) and/or enfuvirtide (ENF).
Drug: Enfuvirtide (ENF) — Participants will receive 2 additonal approved antiretrovirals (ARVs) along with ETR. ARVs may be NRTIs and/or allowed protease inhibitors (PIs) and/or enfuvirtide (ENF).

SUMMARY:
The purpose of this study is to evaluate the long-term safety and tolerability of etravirine, administered as part of an individually optimized antiretroviral therapy (ART), in human immunodeficiency virus Type 1 (HIV-1) infected participants.

DETAILED DESCRIPTION:
This is a Phase II, open-label (all people know the identity of the intervention), roll-over study (participants may go ahead and participate in another clinical study). Participants who were randomized (study medication is assigned by chance) to a etravirine (ETR) treatment arm in Phase II TMC125 feeder studies (TMC125-C203, TMC125-C209, TMC125-C223 and TMC125-C211), were treated for at least 48 weeks with etravirine, and who will derive continued benefit from etravirine therapy, as judged by the investigator, will be enrolled in this study. The final visit of the sponsor-selected Phase II ETR study will be the first (baseline) visit of this study. Approximately 300 participants will be enrolled in this study who will receive 800 mg twice daily of etravirine (formulation TF035) until the formulation 200 mg twice daily (formulation F060) is available. Once this formulation becomes available all the participants will be switched to receive F060 which will be given in combination with an investigator-selected, optimized underlying therapy (nucleotide reverse transcriptase [NRTIs] and/or allowed protease inhibitors and/or enfuvirtide). Participants will continue to receive ETR until they are no longer benefitted or this medication becomes commercially available. Safety evaluations will include assessment of adverse events, clinical laboratory tests, electrocardiogram, vital signs, and physical examination.

ELIGIBILITY:
Inclusion Criteria:

* Participants who were previously randomized to an etravirine (ETR) treatment arm and have completed at least 48 weeks of treatment with ETR
* Participants who will be able to comply with the protocol requirements
* Participants general medical condition should not interfere with the assessments and the completion of the study

Exclusion Criteria:

* Use of disallowed concomitant therapy unless a prior exemption had been granted
* Participant with any treatment-emergent condition or exacerbation of underlying condition during original Phase II study
* Agrees to protocol-defined use of effective contraception
* Participant with a grade 3 elevation of amylase and/or lipase except for isolated grade 3 increases of amylase with lipase in normal range and no history of pancreatitis
* Participant with any grade 4 toxicity according to the Division of Acquired Immunodeficiency Syndrome (DAIDS) grading table; with the exception of grade 4 elevations of triglycerides or glucose asymptomatic or under non-fasting conditions; grade 4 elevation of glucose in participants with pre-existing diabetes
* Participants with clinical or laboratory evidence of significantly decreased hepatic function or decompensation, irrespective of liver enzyme levels (International Normalized Ratio [INR] more than 1.5 or albumin less than 30g/l or bilirubin more than 2.5 x upper limit of normal)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2005-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals, Ireland Clinical Trial, Study Director — Tibotec Pharmaceuticals, Ireland

REFERENCES:
- See also: TMC125-C229: TMC125 in HIV-1 Infected Subjects, Who Were Randomized to a TMC125 Treatment Arm in a Sponsor Selected TMC125 Trial and Were Treated for at Least 48 Weeks — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=980&filename=CR002731_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this study, 211 participants were enrolled in 12 different countries. The majority of participants (49%) were enrolled in the United States.
Pre-assignment Details: In total, 211 participants (93 who rolled over from the etravirine arm of study TMC125-C203 (NCT00412646), 85 who rolled over from the etravirine arm of study TMC125-C223 (NCT00081978), 29 who rolled over from study TMC125-C211 (NCT00111280) and 4 who rolled over from study TMC125-C209) received treatment with etravirine.
Groups:
- Etravirine: 800 mg twice daily (formulation TF035), and after formulation switch, 200 mg twice daily (formulation F060)
Period: Overall Study
Arm/Group | Etravirine
Started | 211
Completed | 139
Not Completed | 72
Not completed — Adverse Event | 10
Not completed — Withdrawal by Subject | 14
Not completed — Lost to Follow-up | 4
Not completed — Reached a virologic endpoint | 29
Not completed — Non-compliant | 4
Not completed — Discontinued or ineligible for study | 2
Not completed — Other | 9

BASELINE CHARACTERISTICS:
Arm/Group | Etravirine
Number analyzed (Participants) | 211
Age Continuous [Median (Full Range); unit: years] | 46.0 (7.56) [32 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 190
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 1
  Black or African American | 24
  White | 164
  Hispanic | 16
  Other | 6

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants Who Achieved Virologic Response (ie, Viral Load Less Than 50 Copies/mL) at Week 48
Description: Number of participants who had viral load more than or equal to 50 copies/mL and less than 50 copies/mL at TMC125-C229 baseline and who achieved virologic response (ie, viral load less than 50 copies/mL) at Week 48. The last visit of the TMC125 feeder study (TMC125-C203 [NCT00412646], TMC125-C223 [NCT00081978], TMC125 C211 [NCT00111280] or TMC125-C209 feeder studies) was considered to be the TMC125-C229 baseline.
Time Frame: Week 48
Population: Intent-to-treat participants who received at least one dose of study medication with evaluable data at Week 48
Measure: Number; unit: Participants
Groups:
- Viral Load More Than or Equal to 50 Copies/mL: Viral load more than or equal to 50 copies/mL at TMC125-C229 Baseline
- Viral Load Less Than 50 Copies/mL: Viral load less than 50 copies/mL at TMC125-C229 Baseline
Arm/Group | Viral Load More Than or Equal to 50 Copies/mL | Viral Load Less Than 50 Copies/mL
Number analyzed (Participants) | 80 | 93
Participants | 22 | 80

2. Secondary Outcome: Number of Participants Who Achieved Virologic Response (ie, Viral Load Less Than 50 Copies/mL) at Week 96
Description: Number of participants who had viral load more than or equal to 50 copies/mL and less than 50 copies/mL at TMC125-C229 baseline and who achieved virologic response (ie, viral load less than 50 copies/mL) at Week 96. The last visit of the TMC125 feeder study (TMC125-C203 [NCT00412646], TMC125-C223 [NCT00081978], TMC125 C211 [NCT00111280] or TMC125-C209 feeder studies) was considered to be the TMC125-C229 baseline.
Time Frame: Week 96
Population: Intent-to-treat participants who received at least one dose of study medication with evaluable data at Week 96
Measure: Number; unit: Participants
Arm/Group | Viral Load More Than or Equal to 50 Copies/mL | Viral Load Less Than 50 Copies/mL
Number analyzed (Participants) | 62 | 83
Participants | 28 | 72

3. Secondary Outcome: Number of Participants Who Achieved Virologic Response (ie, Viral Load Less Than 50 Copies/mL; Less Than 400 Copies/mL; and Greater Than or Equal to 1 Log 10 Decrease From Baseline) at Week 96
Description: Baseline considered for this outcome is the baseline in the respective TMC125-C229 feeder study (TMC125-C203 [NCT00412646], TMC125-C223 [NCT00081978], TMC125 C211 [NCT00111280] or TMC125-C209 feeder studies).
Time Frame: Week 96
Population: Intent-to-treat participants who received at least one dose of study medication with evaluable data at Week 96
Measure: Number; unit: Participants
Arm/Group | Etravirine
Number analyzed (Participants) | 181
Participants
  Viral load (VL) less than 50 copies/mL | 105
  Viral load less than 400 copies/mL | 124
  Viral load more than or equal to 1log10 | 132

4. Secondary Outcome: Number of Participants Who Achieved Virologic Response (ie, Viral Load Less Than 50 Copies/mL; Viral Load Less Than 400 Copies/mL; and Greater Than or Equal to 1 log10 Decrease From Baseline) at Week 192
Description: as for outcome 3
Time Frame: Week 192
Population: Intent-to-treat participants who received at least one dose of study medication with evaluable data at Week 192
Measure: Number; unit: Participants
Arm/Group | Etravirine
Number analyzed (Participants) | 98
Participants
  Viral load (VL) less than 50 copies/mL | 69
  VL less than 400 copies/mL | 81
  VL greater than or equal to 1log10 | 83

5. Secondary Outcome: Median Change From TMC125-C229 Basline in Cluster of Differentiation 4 (CD4+) Cell Count at Week 48
Description: The last visit of the TMC125 feeder study (TMC125-C203 [NCT00412646], TMC125-C223 [NCT00081978], TMC125 C211 [NCT00111280] or TMC125-C209 feeder studies) was considered to be the TMC125-C229 baseline.
Time Frame: Week 48
Population: Intent-to-treat participants who received at least one dose of study medication with evaluable data at Week 48
Measure: Median (Full Range); unit: x 100000 cells/L
Arm/Group | Etravirine
Number analyzed (Participants) | 172
x 100000 cells/L | 21.50 [-422.0 to 1119.0]

6. Secondary Outcome: Median Change From TMC125-C229 Baseline in Cluster of Differentiation 4 (CD4+) Cell Count at Week 96
Description: as for outcome 5
Time Frame: Week 96
Population: Intent-to-treat participants who received at least one dose of study medication with evaluable data at Week 96
Measure: Median (Full Range); unit: x 1000000 cells/L
Arm/Group | Etravirine
Number analyzed (Participants) | 142
x 1000000 cells/L | 18.50 [-460.0 to 391.0]

7. Secondary Outcome: Median Change in Cluster of Differentiation 4 (CD4+) Cell Count From Baseline in TMC125-C229 Feeder Study at Week 96
Description: as for outcome 3
Time Frame: Week 96
Population: Intent-to-treat participants who received at least one dose of study medication with evaluable data at Week 96
Measure: Median (Full Range); unit: x 1000000 cells/mL
Arm/Group | Etravirine
Number analyzed (Participants) | 181
x 1000000 cells/mL | 120.00 [-393.0 to 1590.0]

8. Secondary Outcome: Median Change in Cluster of Differentiation 4 (CD4+) Cell Count From Baseline in TMC125-C229 Feeder Study at Week 192
Description: as for outcome 3
Time Frame: Week 192
Population: Intent-to-treat participants who received at least one dose of study medication with evaluable data at Week 192
Measure: Median (Full Range); unit: x 1000000 cells/mL
Arm/Group | Etravirine
Number analyzed (Participants) | 96
x 1000000 cells/mL | 149.50 [-535.0 to 1847.0]

9. Secondary Outcome: Number of Participants With Emerging Mutation (Reverse Transcriptase Mutation)
Description: Emerging mutations are the mutation which are not present at baseline (last visit of the TMC125 feeder study [TMC125-C203 (NCT00412646), TMC125-C223 (NCT00081978), TMC125 C211 (NCT00111280) or TMC125-C209 feeder studies]) and are present at endpoint (last available timepoint during treatment period for each individual participant).
Time Frame: Baseline and Endpoint (ie, the last available time point during the treatment period)
Population: Intent-to-treat population: Participants who received at least 1 dose of study medication were included
Measure: Number; unit: Participants
Arm/Group | Etravirine
Number analyzed (Participants) | 211
Participants
  L100I | 8
  Y181C | 7
  A98G | 6
  V179I | 6
  K103N | 5
  H221Y | 5

10. Primary Outcome: Number of Participants With Adverse Events
Description: Number of participants who reported at least 1 of the adverse events.
Time Frame: Up to 3 years
Population: Intent-to-treat population: Participants who received at least 1 dose of study medication were included
Measure: Number; unit: Participants
Arm/Group | Etravirine
Number analyzed (Participants) | 211
Participants | 195

ADVERSE EVENTS:
Time Frame: Up to 3 years
Arm/Group | Etravirine
Serious Adverse Events (participants affected / at risk) | 46/211
Other Adverse Events (participants affected / at risk) | 147/211
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etravirine (N=211)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Cardiogenic shock (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Coronary artery occlusion (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 2
Myocardial ischaemia (Cardiac disorders) | 1
Fanconi syndrome (Congenital, familial and genetic disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
Pancreatitis (Gastrointestinal disorders) | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Chest discomfort (General disorders) | 1
Chills (General disorders) | 1
Pyrexia (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Acute sinusitis (Infections and infestations) | 1
Arthritis bacterial (Infections and infestations) | 1
Arthritis infective (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 3
Gastrointestinal infection (Infections and infestations) | 1
Groin abscess (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Histoplasmosis disseminated (Infections and infestations) | 1
Meningitis aseptic (Infections and infestations) | 1
Pneumocystis jiroveCI pneumonia (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 5
Pneumonia viral (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Secondary syphilis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Staphylococcal abscess (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Injury (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Traumatic brain injury (Injury, poisoning and procedural complications) | 1
Biopsy kidney (Investigations) | 1
Biopsy liver (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Diabetes mellitus non-insulin-dependent (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Anal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gum neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Renal artery occlusion (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 2
Renal impairment (Renal and urinary disorders) | 1
Prostatitis (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Abdominoplasty (Surgical and medical procedures) | 1
Hospitalisation (Surgical and medical procedures) | 1
Wound treatment (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Etravirine (N=211)
Lymphadenopathy (Blood and lymphatic system disorders) | 22
Abdominal pain (Gastrointestinal disorders) | 16
Diarrhoea (Gastrointestinal disorders) | 37
Nausea (Gastrointestinal disorders) | 18
Vomiting (Gastrointestinal disorders) | 11
Fatigue (General disorders) | 23
Injection site reaction (General disorders) | 15
Pyrexia (General disorders) | 16
Bronchitis (Infections and infestations) | 15
Nasopharyngitis (Infections and infestations) | 23
Sinusitis (Infections and infestations) | 24
Upper respiratory tract infection (Infections and infestations) | 36
Arthralgia (Musculoskeletal and connective tissue disorders) | 23
Back pain (Musculoskeletal and connective tissue disorders) | 19
Myalgia (Musculoskeletal and connective tissue disorders) | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13
Headache (Nervous system disorders) | 20
Depression (Psychiatric disorders) | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 20
Rash (Skin and subcutaneous tissue disorders) | 16
Hypertension (Vascular disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days